CLINICAL TRIAL: NCT05497349
Title: Use of Leukocyte-Rich PRP or Leukocyte-Free PRP in the Treatment of Hip Osteoarthritis. Double-blind Controlled Randomized Clinical Trial
Brief Title: Use of Leukocyte-Rich PRP or Leukocyte-Free PRP in the Treatment of Hip Osteoarthritis
Acronym: PRP22-Hip
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP22-Hip
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hip Osteoarthritis
Keywords: PRP; LR-PRP; LP-PRP; Platelet rich plasma; PRP injection; Leukocyte Rich-PRP; Leukocyte Poor-PRP; Hip-OA; Hip Osteoarthritis; Randomized controlled trial; Injection treatment
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: The study is a double-blinded RCT in which one group of patients will be treated with 3 intra-articular injection of Leukocyte Rich-PRP, and one group will be treated with 3 intra-articular injection of Leukocyte Poor- PRP
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind randomized controlled trial with allocation 1:1. Patient blinding will be provided during the injection treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leukocyte Rich-PRP Injection (Experimental): Three infiltrations of Leukocyte Rich Platelet Rich Plasma
  1 infiltration weekly, for 3 weeks
  Interventions: Other: Leukocyte Rich- PRP injection
- Leukocyte Poor- PRP Injection (Active Comparator): Three infiltrations of Leukocyte Poor-Platelet Rich Plasma
  1 infiltration weekly, for 3 weeks.
  Interventions: Other: Leukocyte Poor- PRP injection

INTERVENTIONS:
Other: Leukocyte Rich- PRP injection — Autologous Leukocyte Rich-Platelet Rich Plasma will be injected in the hip joint
  Arms: Leukocyte Rich-PRP Injection
Other: Leukocyte Poor- PRP injection — Autologous Leukocyte Poor-Platelet Rich Plasma will be injected in the hip joint
  Arms: Leukocyte Poor- PRP Injection

SUMMARY:
The aim of the study is to compare the efficacy up to 12 months of two different types of PRP (PRP with leukocytes vs PRP depleted of leukocytes) in the echo-guided infiltrative treatment of hip OA by including 230 patients in the study and evaluating them through subjective (using the WOMAC score as the primary outcome) and objective clinical scores.

DETAILED DESCRIPTION:
Platelet-rich plasma (PRP) has recently emerged as an attractive biological approach to address joint degeneration. It has gained increasing attention because of the high concentration of growth factors, cytokines, and bioactive molecules stored in platelet-rich α-granules, which have been shown to participate in joint tissue homeostasis, being involved in both healing processes and immunoregulation and modulation of inflammation. Several preparation methods are available for PRP, which can give products with different compositions and characteristics.The presence of leukocytes is one of the most debated aspects of PRP efficacy, and is used as one of the main discriminators to distinguish different PRPs.

Patients with OA of the hip will be included in a randomized controlled, double-blind trial, in which one group of patients will be treated with 3 infiltrations of PRP with leukocytes and one group will be treated instead with 3 infiltrations of PRP without leukocytes. A total of 230 patients will be included and will undergo infiltrative treatment after collecting informed consent for study participation. Patients will be clinically evaluated before the injection procedure and at 2-6-12 months after treatment by the medical staff.

ELIGIBILITY:
Inclusion Criteria:

* Signs and symptoms of hip OA (pain intensity of at least 4 points and not more than 8 of VAS pain - 0-10 scale in the previous week);
* Radiographic signs of hip OA (Grade 1-2 according to Tonnis classification) or MRI signs (chondropathy or minimal labrum degeneration without acute lesions) even if Grade 0.
* Unilateral involvement; Hemoglobin > 11 g/dl;
* Platelet count > 150,000 plt/mm3 (Recently performed CBC examination);
* Negative serological tests for HBsAg, HCV Ab, HIV-1-2 Ab
* No clinically significant electrocardiographic changes (Recently performed ECG).
* Ability and consent of patients to actively participate in clinical follow-up;- Signature of informed consent.

Exclusion Criteria:

* Patients unable to express consent;
* Patients undergoing infiltration of other substance in the previous 6 months;
* Patients undergoing lower limb surgery to be treated in the previous 12 months;
* Patients with malignant neoplasms;
* Patients with rheumatic diseases;- Patients with uncontrolled diabetes;-Patients with hematological diseases (coagulopathies);
* Patients on anticoagulant-antiaggregant therapy that cannot be discontinued for at least 3 days prior to blood collection;
* Patients with uncontrolled thyroid metabolic disorders;
* Patients abusing alcoholic beverages, drugs or medications;
* Body Mass Index > 30;
* Patients who have taken NSAIDs in the 3 days prior to blood draw;
* Patients with cardiovascular disease for whom 300 ml blood draw would be contraindicated;
* Patients with recently performed CBC examination with Hb< 11 g/dl and Platelet values < 150,000 plt/mm3.
* Positive serological tests for HBsAg, HCV Ab, HIV-1-2 Ab
* Pregnant and/or fertile women.
* Pain intensity less than 4 points or greater than 8 in accordance with the VAS scale.
* Patients with other hip pathologies: acetabular protrusion, concentric migration of the femoral head, presence of excessive deformity resulting from acetabular or femoral head dysplasia, collapse deformity, and deformed femoral head sequelae of Perthes disease or osteonecrosis of the femoral head.
* Previous extensive surgery of the reference joint (osteotomy around the hip, open or arthroscopic osteochondroplasty for femoro-acetabular conflict).

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months follow-up
  It's a standardized and widely used questionnaire to assess the condition of patients with osteoarthritis of the knee and includes assessment of pain, stiffness, and physical function of the joints. It can be administered to the patient.
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); The score is then normalized on a 0-100 scale. Higher values indicate a worse outcome

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline, 2 month and 12 months
  It's a standardized and widely used questionnaire to assess the condition of patients with osteoarthritis of the knee and includes assessment of pain, stiffness, and physical function of the joints. It can be administered to the patient.
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); The score is then normalized on a 0-100 scale. Higher values indicate a worse outcome
Visual Analogue Scale (VAS) | baseline, 2 months, 6 months and 12 months follow-up
  VAS is a visual analogue scale consisting of a range scale (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable".
Harris Hip Scale (HHS) | baseline, 2 months, 6 months and 12 months follow-up
  This scale was developed for the evaluation of hip surgery outcomes and is intended to assess various hip disabilities and treatment methods in an adult population. The four sections that make up the questionnaire are: pain, function, absence of deformity, and range of motion. The HHS is a measure of dysfunction, so higher is the score, better is the outcome for the individual. The maximum possible score is 100.
EQ-5D (EuroQoL) Current Health Assessment | baseline, 2 months, 6 months and 12 months follow-up
  EQ-5D is a standardized measure of health-related quality of life developed by the EuroQol Group to provide a simple generic questionnaire for use in clinical and economic evaluation and population health surveys
Patient Acceptable Symptom State (PASS) | baseline, 2 months, 6 months and 12 months follow-up
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.

CONTACTS AND LOCATIONS:
Overall Officials: Dante Dallari, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Mobasheri A, Batt M. An update on the pathophysiology of osteoarthritis. Ann Phys Rehabil Med. 2016 Dec;59(5-6):333-339. doi: 10.1016/j.rehab.2016.07.004. Epub 2016 Aug 18. PMID 27546496
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Fu M, Zhou H, Li Y, Jin H, Liu X. Global, regional, and national burdens of hip osteoarthritis from 1990 to 2019: estimates from the 2019 Global Burden of Disease Study. Arthritis Res Ther. 2022 Jan 3;24(1):8. doi: 10.1186/s13075-021-02705-6. PMID 34980239
- [Background] Boffa A, Salerno M, Merli G, De Girolamo L, Laver L, Magalon J, Sanchez M, Tischer T, Filardo G. Platelet-rich plasma injections induce disease-modifying effects in the treatment of osteoarthritis in animal models. Knee Surg Sports Traumatol Arthrosc. 2021 Dec;29(12):4100-4121. doi: 10.1007/s00167-021-06659-9. Epub 2021 Aug 2. PMID 34341845
- [Background] Dallari D, Stagni C, Rani N, Sabbioni G, Pelotti P, Torricelli P, Tschon M, Giavaresi G. Ultrasound-Guided Injection of Platelet-Rich Plasma and Hyaluronic Acid, Separately and in Combination, for Hip Osteoarthritis: A Randomized Controlled Study. Am J Sports Med. 2016 Mar;44(3):664-71. doi: 10.1177/0363546515620383. Epub 2016 Jan 21. PMID 26797697
- [Background] Kon E, Mandelbaum B, Buda R, Filardo G, Delcogliano M, Timoncini A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma intra-articular injection versus hyaluronic acid viscosupplementation as treatments for cartilage pathology: from early degeneration to osteoarthritis. Arthroscopy. 2011 Nov;27(11):1490-501. doi: 10.1016/j.arthro.2011.05.011. Epub 2011 Aug 10. PMID 21831567
- [Background] Ornetti P, Nourissat G, Berenbaum F, Sellam J, Richette P, Chevalier X; under the aegis of the Osteoarthritis Section of the French Society for Rheumatology (Societe Francaise de Rhumatologie, SFR). Does platelet-rich plasma have a role in the treatment of osteoarthritis? Joint Bone Spine. 2016 Jan;83(1):31-6. doi: 10.1016/j.jbspin.2015.05.002. Epub 2015 Jul 7. PMID 26162636
- [Background] Battaglia M, Guaraldi F, Vannini F, Rossi G, Timoncini A, Buda R, Giannini S. Efficacy of ultrasound-guided intra-articular injections of platelet-rich plasma versus hyaluronic acid for hip osteoarthritis. Orthopedics. 2013 Dec;36(12):e1501-8. doi: 10.3928/01477447-20131120-13. PMID 24579221
- [Background] Di Sante L, Villani C, Santilli V, Valeo M, Bologna E, Imparato L, Paoloni M, Iagnocco A. Intra-articular hyaluronic acid vs platelet-rich plasma in the treatment of hip osteoarthritis. Med Ultrason. 2016 Dec 5;18(4):463-468. doi: 10.11152/mu-874. PMID 27981279
- [Background] Ye Y, Zhou X, Mao S, Zhang J, Lin B. Platelet rich plasma versus hyaluronic acid in patients with hip osteoarthritis: A meta-analysis of randomized controlled trials. Int J Surg. 2018 May;53:279-287. doi: 10.1016/j.ijsu.2018.03.078. Epub 2018 Apr 5. PMID 29626641
- [Background] Di Martino A, Boffa A, Andriolo L, Romandini I, Altamura SA, Cenacchi A, Roverini V, Zaffagnini S, Filardo G. Leukocyte-Rich versus Leukocyte-Poor Platelet-Rich Plasma for the Treatment of Knee Osteoarthritis: A Double-Blind Randomized Trial. Am J Sports Med. 2022 Mar;50(3):609-617. doi: 10.1177/03635465211064303. Epub 2022 Feb 1. PMID 35103547
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365